CLINICAL TRIAL: NCT01896583
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Pilot Study to Assess the Efficacy, Safety and Tolerability, of ASP7147 in Patients With Diarrhea Predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: A Phase 2 Pilot Study to Assess ASP7147 in Patients With Diarrhea Predominant Irritable Bowel Syndrome (IBS-D)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seldar Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7147-CL-0003
Record Dates: First submitted 2013-06-26; First posted 2013-07-11 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Diarrhea Predominant Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- ASP7147 (Experimental): ASP7147, 300 mg, tablet, twice per day for 4 weeks oral
  Interventions: Drug: ASP7147
- Placebo (Placebo Comparator): oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP7147 — 300 mg, tablet, twice per day for 4 weeks oral
  Arms: ASP7147
Drug: Placebo
  Arms: Placebo

SUMMARY:
This trial will evaluate the effect of ASP7147 on daily abdominal pain due to IBS-D during 4 weeks of treatment. It will also evaluate safety and tolerability in patients with IBS-D over the 4-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Men or women aged 18-75 years
* Patient has IBS with diarrhea (IBS-D)
* Ability to communicate with the investigator

Exclusion Criteria:

* IBS with constipation (IBS-C) or mixed IBS (IBS-M)
* Other significant disease or condition that may interfere with trial completion
* Untreated lactose intolerance
* History of alcohol or drug abuse in past two years
* Participation in other clinical trials within prior month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Abdominal pain | 4 weeks
  10-point pain scale

SECONDARY OUTCOMES:
Stool consistency | 4 weeks
  Bristol Stool Scale (7-point scale)
Stool frequency | 4 weeks
  Number of bowel movements per day

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Elite Clinical Studies, Phoenix, Arizona
  - Shahram Jacobs, M.D., Inc., Encino, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - Probe Clinical Research Group, Santa Ana, California
  - San Marcus Research Clinic Inc, Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Meridien Research, St. Petersburg, Florida
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Sundance Clinical Research, St Louis, Missouri
  - OM Medical, Las Vegas, Nevada
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Remington-Davis, Inc., Columbus, Ohio
  - DCT - Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas